CLINICAL TRIAL: NCT04974424
Title: Study on Early Warning Model of Susceptibility and High-risk Population of Cervical Cancer Related to HPV
Brief Title: Early Warning Model of Susceptibility and High-risk Population of Cervical Cancer Related to HPV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Women's Hospital School Of Medicine Zhejiang University (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Qilu Hospital of Shandong University (Other); Wuhan Central Hospital (Other); Third Military Medical University (Other); Xiangyang Central Hospital (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Principal Investigator, Ding Ma, Director of Obstetrics and Gynecology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: S160
Record Dates: First submitted 2021-06-24; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Uterine Cervical Neoplasm; Uterine Cervical Cancer; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Most uterine cervical high-risk human papillomavirus (HPV) infections are transient, with only a small fraction developing into cervical cancer. Family aggregation studies and heritability estimates suggest a significant inherited genetic component. Candidate gene studies and previous genome-wide association studies (GWASs) report associations between the HLA region and cervical cancer. Adopting a genome-wide approach, we aimed to establish an early warning model for a high-risk population of cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Case group a) Aged 25-75 years. b) Han nationality. c) Patients with cervical cancer or cervical precancerous lesions above CIN2 diagnosed by biopsy or postoperative pathological diagnosis.
* (2) Control group: a) Aged 25-75 years. b) Han nationality. c) No family history of cervical cancer or precancerous lesions. d) The results of TCT examination showed no abnormality.

Exclusion Criteria:

* (1) suffering from other neoplastic diseases.
* (2) pregnant women.
* (3) those with a history of bone marrow transplantation.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese population
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Significant loci of genetic variation | 2
  The impact of genetic variance on predisposition to cervical cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, MD, PhD, Study Chair — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China